CLINICAL TRIAL: NCT02494492
Title: Treatment of the Bilateral Severe Uveitis by IVT of Regulator T-cells: Study of Tolerance of Dose
Acronym: UVEREG
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P081250
Record Dates: First submitted 2015-06-10; First posted 2015-07-10 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Uveitis
Keywords: Uveitis; Lymphocyte cells; lymphocyte T regulator; vitreous haze; intravitreal injection
MeSH Terms: conditions — Uveitis | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVT of regulator T-cells (Experimental): intravitreous administration of regulator T-cells
  Interventions: Other: intravitreous administration of regulator T-cells

INTERVENTIONS:
Other: intravitreous administration of regulator T-cells — The 3 levels of Tregs doses will be respectively 0.4, 1.2 and 3.6 million.
  Other Names: cell therapy

SUMMARY:
Uveitis is a leading cause of blindness in the children and young adult's populations. One third of etiology are idiopathic. The reference treatments are corticosteroids and immunosuppressive agents. They have significant side effects, and patient's compliance is often poor. In addition, some uveitis are more resistant. Also, in these situations of deadlock therapeutic, investigators propose a cell therapy by administering regulatory T cells (Tregs) in the vitreous of patients.

DETAILED DESCRIPTION:
Arsenal and limitations in the treatment of uveitis Uveitis is a major cause of severe visual loss or even blindness in children and young adults. In almost one third of cases, it is associated with an infectious agent, another third is integrated in the field of autoimmune diseases as systemic entities including (Behçet's disease, sarcoidosis, spondyloarthropathy ...) or limited to the eye (Birdshot type retinochoroidopathy, sympathetic ophthalmia, idiopathic retinal vasculitis). The last third remains idiopathic, where despite a careful etiological research, no cause is identified. The systemic corticosteroids are often effective but have significant side effects and patient compliance is often poor. That is why they are sometimes administered directly into the posterior segment of the eye (vitreous), but the effect is only temporary, often ineffective, and also associated with side effects. In addition, some are steroid-dependent, requiring treatment with immunosuppressive agents; which also may be responsible for many adverse effects and are not always effective. In these therapeutic impasse situations, investigators propose a cell therapy approach injection of CD4 + CD25 + Foxp3 regulators + (Tregs), directly into the vitreous of patients.

A new therapy approach uveitis by cell therapy It is now clearly established that Tregs play a critical role in the control of autoimmune diseases. In man or mouse, a deep deficit in Tregs is associated with a very severe autoimmune syndrome, leading to death .In uveitis, it is also shown that Tregs control this disease in deficient mice. Tregs have been reported in humans . In addition, our group and others have shown that various autoimmune diseases can be prevented by transfer of Tregs in mice .Thus, cell therapy by injection of Tregs raises hopes for the treatment of chronic inflammatory and autoimmune diseases . However, only specific and not polyclonal Tregs, have a strong therapeutic potential when administered systemically. The only Tregs that can be used in clinic are polyclonal Tregs purified by magnetic beads to which, are adsorbed anti- CD25 antibody . This technology provides a cell preparation enriched in Tregs for 50 to 70%, the balance consisting of effector T cells (Teffs ) , B lymphocytes and NK cells. A therapeutic alternative to the systemic injection of specific Tregs is to inject, preactivated polyclonal Tregs directly into the target site of autoimmune disease, in purified clinical grade condition.

Description of the study population. Patients with bilateral severe steroid-dependent non-infectious uveitis. Infectious or tumoral etiologies have been excluded after completion of a comprehensive review of systems. All patients had a negative Quantiferon test and a normal Mantoux test. Biological tests sent to specialized laboratories will eliminate an active infection. In some cases, aqueous humor obtained after AC tap and / or vitreous biopsy obtained after vitrectomy will be analyzed for diagnostic assay IL-10, immune load factor or PCR analysis (toxoplasmosis, herpes viruses).

Pathophysiology of uveitis in humans. Inflammatory chemokines and cytokines, such as IL-6, IFN-g, IL-8 and MCP-1 and sometimes IL-1ß, IL-2 and TNF-alpha were found in the aqueous humor and vitreous of patients with uveitis . Given the small volume available in these human samples (around 100 ml), data are obtained with multiple detection techniques using flow cytometry, for measuring the concentration of thirty different cytokines and chemokines in a 50 microl volume.

In order to expand the study to other cytokines and chemokines, investigators also used a semi-quantitative technique named ""antibody array"" which allows the analysis of a number of different molecules ranging from 30 to 170. These preliminary results, evaluated in some patients, confirm the presence of Th1 inflammatory profile in the eye of patients suffering from uveitis (not shown) and confirm our strategy

Risks associated with injected cells. No side effects of Tregs injection has been observed in preclinical mouse model. In our Biotherapies facilities, production of Tregs, as provided in this essay, will contain 50 to 70% of Tregs, defined by the phenotype CD4 + Foxp3 + CD25 +. Therefore investigators tested the effect of leukocyte contaminants on therapeutic effect in uveitis in mice. The presence of such contaminants effector T cells, B cells, NK cells, dendritic cells or macrophages did not cause visible side effects at the clinical or histological levels. A second potential risk is that the injected of polyclonal Tregs have been differentiated into a different celltype. Anterior study showed that natural human Tregs can differentiate into Th17 type T lymphocytes in the presence of IL-2 or IL-15. This differentiation is accentuated by the addition of IL-1ß, IL-6, IL-21 or IL-23 . Although investigators can not formally exclude the possibility that Tregs injected IVT may differentiate into Th17 cells, since this event is not probably been detected in uveitis eye (data not shown).

Another potential risk of dissemination of the injected cells from the eye due to reflux at conjunctiva during the IVT. The last risk that can be considered is the development of non- Hodgkin lymphoma by creating a tolerogenic environment due to regulatory T cells. This risk is identical than the one associated with the current reference treatment of uveitis : immunosuppressives agent and corticosteroids. These risks have never been fully described in the literature in both animals and humans.

Dosage and number of patients. The 3 levels of Tregs doses will be respectively 0.4, 1.2 and 3.6 million. The lowest dose of 0.4 million Tregs corresponding to 2 times the effective dose in mice.

Two to 18 patients will be enrolled in this trial. Funding is provided for 12 patients.

Good clinical practice( GCP) The research will be conducted in accordance with GCP and the current legislative and regulation. Investigators certify that the research will be conducted in accordance with the protocol of GCP The Biotherapies facilities perform production activities, quality control according to current regulations for cell therapy and compliance with good practices of Cellular Therapy (BPTC) and also according to standard operating procedures (SOP). Specific authorization is required from ANSM for the realization of this essay To conclude, it is now clearly established that cell therapy approach of CD4 + CD25 + Foxp3 regulators (Tregs) play a critical role in the control of autoimmune diseases in human or mouse clinical test . Therefore this clinical trial assess the effect of Tolerance- dose of in patients treated by Tregs for bilateral severe steroid-dependent non-infectious uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years
* severe bilateral uveitis not infectious
* visual acuity between CLD and 1/10 for the eye the most affected and less than 5/10 for the fellow eye
* failed steroid ≤ 15 mg / day with or without an immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity (occurrence of at least 2 ocular serious adverse events) | 4 weeks
  Toxicity (or intolerance) is defined as the occurrence of at least 2 ocular serious adverse events in 4 weeks following the injection of
  Treg, defined as:
  * an increase on OCT of the retinal thickness of <800mm from the initial review of the visit 1 of the eye injected,
  * decrease in visual acuity compared to the initial review of the visit 1of the eye injected with 2 lines,
  * occurence of ocular hypertension uncontrolled by ≥ 21 mmHg local treatment or hypotonia (5mmHg) compared to the initial review of the visit 1 of the eye injected,
  * occurence of vitreous hemorrhage, retinal necrosis, except complications attributed to the technique of administration,
  * onset of a hypopyon, except complication attributed to the technical Board

SECONDARY OUTCOMES:
ETDRS scale | 4 weeks
  visual acuity measured by ETDRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Bahram BODAGHI, Professor, Principal Investigator — Assitance publique - Hopitaux de Paris
Locations (1):
- Department of ophthalmology Groupe Hospitalier Pitié-Salpêtrière - Charles FOIX, Paris, France